CLINICAL TRIAL: NCT04600895
Title: Favipiravir for Patients With Mild to Moderate Disease From Novel Coronavirus (COVID-19)
Brief Title: The Prevent Severe COVID-19 (PRESECO) Study
Acronym: PRESECO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Appili Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATI0220
Record Dates: First submitted 2020-09-15; First posted 2020-10-23 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Experimental): Favipiravir 200mg tablet
  Interventions: Drug: Favipiravir
- Placebo (Placebo Comparator): Placebo 200mg tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Favipiravir — Favipiravir
  Arms: Favipiravir
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Double-blinded, placebo control, randomized, phase-3 clinical trial to evaluate clinical efficacy of Favipiravir in patients with mild to moderate symptoms related to COVID-19 infection

DETAILED DESCRIPTION:
COVID-19 starts as a pure viral infection and evolves into a multifactorial disease with components of hyper immune activation, end organ damage, and fibrosis. Suppression of viral replication is expected to be impactful early in the course of disease. The ability to mitigate the symptoms at an early stage will prevent progression to severe COVID-19 and can save many lives. Early treatment could also reduce viral shedding, diminishing the period of infectivity and decreasing the number of secondary cases.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Tested positive for SARS-CoV-2 by RT-PCR assay using a respiratory tract sample (either nasopharyngeal swab OR oropharyngeal swab OR nasal aspirate OR tracheobronchial aspirate OR saliva) collected within 72 hours of randomization
* Stated willingness to give their written informed consent to participate in the study
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Males must be sterile, OR agree not to donate semen AND agree to strictly adhere to contraceptive measures during the study and for 7 days following the last dose of study medication
* Females must be unable to bear children, OR ensure that their male partner is incapable of fathering a child, OR, if of childbearing potential will strictly adhere to contraceptive measures during the study and for seven days following the last dose of study medication
* Females must agree to stop breast-feeding prior to first dose of study drug and through seven days after completing therapy
* Females must have a negative pregnancy test at screening
* Ability to take oral medication and be willing to adhere to the favipiravir/placebo regimen
* Subject has access to a smart phone, tablet, or PC
* Minimal baseline severity score for COVID-19-related symptoms: at least two symptoms with a score of 2 or higher. COVID-19-related symptoms (excluding changes in the sense of taste or smell) include:
* stuffy or runny nose
* sore throat
* shortness of breath
* cough
* lack of energy or tiredness
* muscle or body aches
* headache
* chills or shivering
* feeling hot or feverish
* nausea
* diarrhea
* vomiting

Exclusion Criteria:

* O2 saturation <94%
* Shortness of breath at rest
* Heart rate ≥ 125 per minute
* COVID-19 symptoms first presented >5 days prior to randomization
* Requirement for hospitalization at the time of enrollment
* Participation in another trial or use of any experimental treatment for COVID-19
* Treatment with high steroid dose i.e. >30 mg/day prednisolone equivalent (excluding stable chronic treatment) or remdesivir or anyone receiving SARS-CoV-2 monoclonal antibodies within 3 months prior to enrollment
* Known sepsis or organ dysfunction/ failure
* Known infection with a respiratory virus other than SARS-CoV2 (e.g. Influenza) or any known bacterial infection (affecting the respiratory system or any other system)
* Inability to adhere to study requirements
* For premenopausal women: unwilling or unable to use effective birth control measures
* Known allergy to favipiravir
* Known end-stage kidney disease or requiring hemodialysis or continuous ambulatory peritoneal dialysis (CAPD)
* Known liver impairment greater than Child-Pugh A
* Psychiatric illness that is not well controlled (defined as stable on a regimen for more than one year).
* Known elevated uric acid levels in the past year or taking uric acid lowering medications (allopurinol, febuxostat)
* History of hereditary xanthinuria or history of xanthine urolithiasis.
* History of gout or actively being treated for gout.
* Current use of the following medications, which cannot be discontinued for the duration of the study: pyrazinamide, hydralazine, more than 3000 mg of acetaminophen per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1187 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (25):
  - Cahaba Research, Inc., Pelham, Alabama
  - Absolute Clinical Research, Phoenix, Arizona
  - B.G Clinical Research Center, LLC, Little Rock, Arkansas
  - Xera Med Research, Boca Raton, Florida
  - Synergy Healthcare, Bradenton, Florida
  - Best Quality Research,Inc., Hialeah, Florida
  - Elixia Clinical Research Collaborative, Hollywood, Florida
  - Homestead Associates In Research, Miami, Florida
  - Verus Clinical Research Corporation, Miami, Florida
  - Quality Professional HealthCare, Miami, Florida
  - Continental Clinical Research, LLC, Miami, Florida
  - Global Life Research Network, Llc, Miami, Florida
  - Sanitas Research, LLC, Miami, Florida
  - US Associates in Research, LLC, Miami, Florida
  - Biore'Search Institute Llc, Pembroke Pines, Florida
  - Luminous Clinical Research - South Florida Urgent Care, Pembroke Pines, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - University of Massachusettts Medical School, Worcester, Massachusetts
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - New Phase Research & Development, Knoxville, Tennessee
  - Next Level Urgent Care, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Frontier Clinical Research, Kingwood, West Virginia
- Brazil (7):
  - Centro de Pesquisas Clínicas de Natal, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - LMK Servicos Medicos S/S, Porto Alegre, Rio Grande do Sul
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Pesquisare Saude S/S LTDA, Santo André, São Paulo
  - Centro Medico Mazzei, São Paulo
  - Hospital Santa Paula, São Paulo
- Mexico (6):
  - Invesclinic Mx, Irapuato, Guanajuato
  - Kohler & Milstein Research S.A. de C.V, Yucatán, Merida
  - JM Research SC, Cuernavaca, Morelos
  - Tecsi S.C., Monterrey, Nuevo León
  - Panamerican Clinical Research Mexico, S.A. de C. V., Juriquilla, Querétaro
  - Centro Medico Espiritu Santo, Tequisquiapan, Querétaro

REFERENCES:
- [Derived] Golan Y, Campos JAS, Woolson R, Cilla D, Hanabergh R, Gonzales-Rojas Y, Lopez R, Finberg R, Balboni A. Favipiravir in Patients With Early Mild-to-moderate Coronavirus Disease 2019 (COVID-19): A Randomized Controlled Trial. Clin Infect Dis. 2023 Feb 8;76(3):e10-e17. doi: 10.1093/cid/ciac712. PMID 36065065

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Favipiravir | Placebo
Started | 599 | 588
ITT | 599 | 588
MITT | 599 | 588
MITT2 | 539 | 505
Completed | 480 | 462
Not Completed | 119 | 126

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Favipiravir | Placebo | Total
Number analyzed (Participants) | 599 | 588 | 1187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 543 | 544 | 1087
  >=65 years | 56 | 44 | 100
Age, Continuous [Median (Full Range); unit: years] | 42 [18 to 85] | 44 [18 to 87] | 43 [18 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 317 | 327 | 644
  Male | 282 | 261 | 543
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 63 | 59 | 122
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 43 | 26 | 69
  White | 485 | 491 | 976
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 482 | 480 | 962
  Brazil | 35 | 30 | 65
  Mexico | 82 | 78 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Clinical Recovery
Description: The endpoint will be considered to have been met at the earliest time point at which the subject has reached Sustained Alleviation of Symptoms (Symptoms related to smell or taste are not included in the primary endpoint) reported by the patient have reached a severity of "0 - none" or "1 - mild" in assessments for 4-point scale assessments and not known to have redeveloped any COVID-19 associated signs and symptoms (not including reduced sense of taste or smell) in a severity beyond mild for 4 consecutive days when assessed from the start of study treatment to day 28. To meet the primary endpoint, subjects must survive with no hospitalization to day 28.
Time Frame: From Day 0 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir | Placebo
Number analyzed (Participants) | 599 | 588
Participants | 425 | 475

2. Secondary Outcome: Proportion of Subjects With COVID-19 Progression (Narrow Progression)
Description: Proportion of subjects with COVID-19 progression, where progression is defined as the occurrence from study day 3 onward of any emergency department (ED) visit for COVID-19 worsening or shortness of breath OR hospitalization for COVID-19 worsening or shortness of breath OR death (narrow progression)
Time Frame: From study day 3 to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir | Placebo
Number analyzed (Participants) | 599 | 588
Participants | 174 | 113

ADVERSE EVENTS:
Time Frame: From baseline through Day 28
Arm/Group | Favipiravir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/599 | 1/588
Serious Adverse Events (participants affected / at risk) | 12/599 | 14/588
Other Adverse Events (participants affected / at risk) | 84/599 | 89/588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favipiravir (N=599) | Placebo (N=588)
Covid-19 (Infections and infestations) | 12 (12) | 14 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favipiravir (N=599) | Placebo (N=588)
Nausea (Gastrointestinal disorders) | 8 (8) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 10 (10)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Anosmia (Nervous system disorders) | 1 (1) | 4 (4)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2)
Burning sensation (Nervous system disorders) | 1 (1) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 2 (2)
Hypogeusia (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (21) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (13)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (21) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (21) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (21) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 6 (16) | 5 (17)
Pneumonia (Infections and infestations) | 2 (16) | 5 (17)
COVID-19 (Infections and infestations) | 3 (16) | 3 (17)
Nasopharyngitis (Infections and infestations) | 1 (16) | 1 (17)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (17)
Bronchitis (Infections and infestations) | 0 (0) | 1 (17)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (17)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (17)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (17)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (17)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (17)
Sinusitis (Infections and infestations) | 1 (16) | 0 (0)
Chest discomfort (General disorders) | 4 (11) | 1 (11)
Chest pain (General disorders) | 0 (0) | 3 (11)
Hypothermia (General disorders) | 2 (11) | 1 (11)
Pyrexia (General disorders) | 1 (11) | 2 (11)
Chills (General disorders) | 2 (11) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (11)
Asthenia (General disorders) | 1 (11) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (11)
Malaise (General disorders) | 0 (0) | 1 (11)
Peripheral swelling (General disorders) | 1 (11) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 7 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (6) | 1 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (6) | 1 (11)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (11)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (11)
Rash (Skin and subcutaneous tissue disorders) | 5 (10) | 2 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (10) | 3 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (10) | 1 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (10) | 1 (7)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (10) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (10) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (10) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (7)
Blood uric acid increased (Investigations) | 2 (6) | 0 (0)
Serum ferritin increased (Investigations) | 1 (6) | 1 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (7)
Blood glucose increased (Investigations) | 0 (0) | 1 (7)
Blood potassium increased (Investigations) | 0 (0) | 1 (7)
C-reactive protein increased (Investigations) | 1 (6) | 0 (0)
Electrocardiogram ST-T segment abnormal (Investigations) | 1 (6) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (7)
Heart rate increased (Investigations) | 0 (0) | 1 (7)
Hepatic enzyme increased (Investigations) | 1 (6) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (7)
Liver function test increased (Investigations) | 1 (6) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (4) | 1 (5)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (5) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (5) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (5) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (5) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (5) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 2 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (3)
Restlessness (Psychiatric disorders) | 1 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 1 (3)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (3) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT04600895/Prot_SAP_000.pdf